CLINICAL TRIAL: NCT02799121
Title: A Feasibility Study of the ReGenerCell™ Autologous Cell Harvesting Device for Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP005
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReGenerCell™ (Experimental): Debridement and/or a sterile saline rinse of ulcer, as clinically indicated, followed by ReGenerCell™ treatment and appropriate dressing and off-loading
  Interventions: Device: ReGenerCell™ Autologous Cell Harvesting Device

INTERVENTIONS:
Device: ReGenerCell™ Autologous Cell Harvesting Device

SUMMARY:
This prospective case series is to gain additional clinical experience in the treatment of diabetic foot ulcers, by documenting and relating patient history (including baseline wound characteristics) and clinical outcomes (incidence of healing, rate of healing, and patient and physician satisfaction) in a group of study participants for whom the ReGenerCell™ Autologous Cell Harvesting Device (ReGenerCell™) is used in combination with conventional therapy for the closure of diabetic foot ulcers (DFUs). Participants will receive ReGenerCell™ treatment in addition to standard care (debridement, cleansing, dressings, offloading).

ELIGIBILITY:
Inclusion Criteria:

* The patient has stable diabetes mellitus according to investigators clinical judgement
* Diabetic foot Ulcer

  * Groups 1 and 2: Ulcer surface area between 3 cm2 and 100 cm2 (inclusive)
  * Group 1: 12-24 weeks in duration, no directly visible tendon or bone (University of Texas Ulcer grade 1A)
  * Group 2: >3 weeks in duration, University of Texas Ulcer grade 1B, 2A, 2B, 3A, 3B
* No superficial skin infection (of the ulcer area) requiring intervention
* Adequate offloading and compliance must be achievable
* The patient is 18 years of age or older
* The patient is willing to complete all follow-up evaluations required by the study protocol
* The patient is able to abstain from any other non-standard treatment of the ulcer for the duration of the study, unless medically necessary
* The patient agrees to abstain from enrolment in any other interventional clinical trial for the duration of the study
* The patient is able to read and understand instructions and give voluntary written informed consent
* The patient is able and willing to follow the protocol

Exclusion Criteria:

* Patients requiring intervention for Peripheral Arterial Disease (PAD) will be excluded from this study
* Severe Peripheral Arterial Disease that is not reconstructible
* Pregnant/lactating females (self-reported or tested, per institutional requirements
* Use of non-inert dressings (silver, honey etc.) during the past 10 days
* Subjects who have evidence of connective tissue disorders (e.g. vasculitis or rheumatoid arthritis) under active treatment
* The patient is known to have a pre-existing active condition that may interfere with wound healing, e.g. malignancy, autoimmune disease, immunocompromised blood borne diseases, the patient has AIDS, is HIV- or Hepatitis-C positive, or currently has a severe dermatological disorder (e.g. severe psoriasis, epidermolysis bullosa, pyoderma gangrenosum).
* The patient is taking, or has taken in the past 60 days, >10mg of corticosteroids per day.
* The patient has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives
* The patient has a known hypersensitivity to trypsin or Compound Sodium Lactate solution.
* The patient is a vulnerable or protected adult
* The patient is unable to follow the protocol
* The patient is unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Complete Wound Closure | 26 Weeks
  100% Re-epithelialisation of wound

SECONDARY OUTCOMES:
Wound size | 26 Weeks
  Objectively measured ulcer area cmxcm
Neuro-QoL | 26 Weeks
  Quality of Life short questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - King's College Hospital, London, London
  - Northwick Park Hospital, London
  - Manchester Royal Infirmary, Manchester